CLINICAL TRIAL: NCT04036110
Title: Vitamin C Supplementation Intervention for Patients With Heart Failure-A Pilot Study
Brief Title: Vitamin C Supplementation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-1809; T32NR007091 (NIH)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure
Keywords: Vitamin C supplementation
MeSH Terms: conditions — Heart Failure | interventions — Ascorbic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Experimental): Vitamin C 500 mg taken daily for 3 months
  Interventions: Dietary Supplement: Vitamin C 500 mg
- Intervention 2 (Experimental): Vitamin C 1000 mg taken daily for 3 months
  Interventions: Dietary Supplement: Vitamin C 1000 mg
- Control (Placebo Comparator): Placebo tablets taken daily for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C 500 mg — 500 mg tablet taken orally with one meal daily
  Other Names: L-Ascorbic acid
  Arms: Intervention 1
Dietary Supplement: Vitamin C 1000 mg — 1000 mg tablet taken orally with one meal daily
  Other Names: L-Ascorbic acid
  Arms: Intervention 2
Other: Placebo — 1 tablet taken orally with one meal daily
  Other Names: Sugar pill
  Arms: Control

SUMMARY:
This study is to test a low-cost, simple vitamin C supplementation intervention, that is, comparing placebo to 500 mg/day vitamin C and 1 gram/day vitamin C daily to assess feasibility and acceptability of vitamin C supplementation and effects on serum vitamin C level, health-related quality of life (HRQOL), symptom burden, oxidative stress, and cardiac function.

DETAILED DESCRIPTION:
This study will address feasibility from the perspective of being able to: a) to detect significant differences in the serum vitamin C level after supplementation (3 months) between the intervention groups and the control group, b) to detect significant differences in health related quality of life (HRQOL), symptom burden, oxidative stress, and cardiac function after vitamin C supplementation (3 months) between the intervention groups and the control group.

ELIGIBILITY:
Inclusion Criteria:

Patents recruited will have a diagnosis of chronic HF, either preserved or reduced ejection fraction. The diagnosis and etiology of chronic HF will be confirmed by a HF cardiologist using established criteria.

Other criteria:

* have undergone evaluation of HF and optimization of medical therapy,
* vitamin C supplementation <500 mg/day
* have not been referred for heart transplantation,
* able to read and speak English,
* >1 month from any inpatient hospitalization

Exclusion Criteria:

* history of renal stones or renal disease (serum creatinine >1.5,
* history of glucose-6-phosphate dehydrogenase deficiency (G6PD) and cognitive impairment that precludes giving informed consent or ability to follow protocol instructions
* pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Rong Wu, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNCH Meadowmont Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared, after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication from this trial.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Carr AC, Vissers MC, Cook JS. The effect of intravenous vitamin C on cancer- and chemotherapy-related fatigue and quality of life. Front Oncol. 2014 Oct 16;4:283. doi: 10.3389/fonc.2014.00283. eCollection 2014. PMID 25360419
- [Background] Ellis GR, Anderson RA, Chirkov YY, Morris-Thurgood J, Jackson SK, Lewis MJ, Horowitz JD, Frenneaux MP. Acute effects of vitamin C on platelet responsiveness to nitric oxide donors and endothelial function in patients with chronic heart failure. J Cardiovasc Pharmacol. 2001 May;37(5):564-70. doi: 10.1097/00005344-200105000-00008. PMID 11336107

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study briefly suspended due to administrative reasons.
Groups:
- Intervention 1 (500 mg): Participants take vitamin C (L-Ascorbic acid) 500 mg tablet orally with one meal daily for 3 months
- Intervention 2 (1000 mg): Participants take vitamin C (L-Ascorbic acid) 1000 mg tablet orally with one meal daily for 3 months
- Control (Placebo): Participants take vitamin C placebo (Sugar pill) tablet orally with one meal daily for 3 months
Period: Overall Study
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Started | 12 | 12 | 12
Completed | 5 | 5 | 10
Not Completed | 7 | 7 | 2
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Study Suspended | 4 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 11 | 30
  >=65 years | 4 | 1 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (18) | 51 (14) | 56 (8) | 54 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 9
  Male | 9 | 7 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 8 | 19
  White | 7 | 5 | 4 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Serum Vitamin C Level at Baseline
Description: The ELISA (enzyme-linked immunosorbent assay) used to detect and quantify Vitamin C in serum
Time Frame: Baseline
Population: Data unreported for participants who refused to provide blood sample
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 10 | 10 | 12
ng/mL | 13372 (11555) | 16079 (12564) | 13111 (9135)

2. Primary Outcome: Serum Vitamin C Level at Month 3
Description: The ELISA (enzyme-linked immunosorbent assay) used to detect and quantify Vitamin C in serum
Time Frame: Month 3
Population: Data unreported for participants who refused to provide blood sample
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 2 | 4 | 7
ng/mL | 21309 (11740) | 20574 (13144) | 12537 (7945)

3. Secondary Outcome: Health Related Quality of Life Scores
Description: Health related quality of life is measured using the Minnesota Living with Heart Failure questionnaire (MLHFQ). The MLHFQ is a patient-reported outcome to measure the patient's perceptions of the influence of heart failure on physical and emotional aspects of life. The questionnaire has 21 items to assess the impact of frequent physical symptoms of heart failure and the effects of heart failure on physical and emotional functions. The response scale for all 21 items on the MLHFQ is based on a 6-point (from 0 to 5). Scores are summed to a range of 0-105, in which with higher scores indicate worse health-related quality of life. Measured at Baseline and Month 3.
Time Frame: Baseline and up to 3 months after enrollment
Population: Data unreported for some participants due to study suspended and lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 5 | 5 | 10
score on a scale
  Baseline | 45.3 (32.2) | 31.4 (24.7) | 44.2 (31.4)
  Month 3 | 68.2 (23.2) | 47.4 (37.9) | 27.6 (27.6)

4. Secondary Outcome: Total MSAS-HF Score
Description: Symptom burden is measured using items from the Memorial Symptom Assessment Scale-Heart Failure (MSAS-HF). The MSAS-HF is an 8-item questionnaire to measure HF symptoms experienced by patients with HF. Patients will be first asked if the symptom was present during the previous 7 days. If present, three characteristics of each symptom will be rated: frequency of symptom, severity of symptom, and degree of symptom distress. Frequency is rated on a scale from 0 to 5 (1=no symptom to 5=all the time), severity rated on a scale from 0 to 5 (0=not at all to 5=extremely) and distress rated on a scale from 0 to 5 (0=not at all to 5=extremely). Burden score for each symptom can range from 0 (no burden) to 4 (greatest symptom frequency, severity, and distress). The total MAS-HF scores are summed to a range of 0-180, with higher scores indicating higher symptom burden. Measured at Baseline and Month 3.
Time Frame: Baseline and up to 3 months after enrollment
Population: Data unreported for some participants due to study suspended and lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 5 | 5 | 10
score on a scale
  Baseline | 47.5 (42.7) | 20.2 (26.6) | 31.2 (26.8)
  Month 3 | 24.5 (33.3) | 24.8 (41.4) | 20.1 (30.0)

5. Secondary Outcome: Cardiac Function
Description: The MindWare Mobile impedance cardiograph (model number 50-2303-00) used to measure participant's cardiac function using the parameter of cardiac output. Measured at Baseline and Month 3.
Time Frame: Baseline and up to 3 months after enrollment
Population: Data missing due to staff learning curve using the MindWare Mobile impedance cardiograph and technical problems to detect signal from participants with pacemaker devices which caused inability to measure impedance cardiograph.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 1 | 0 | 2
L/min
  Baseline | 6.9 |  | 5.6 (5.1)
  Month 3 | 12.7 |  | 14.2 (5.1)

6. Secondary Outcome: Oxidative Stress
Description: The ELISA (enzyme-linked immunosorbent assay) used to detect and quantify 8-iso-PGF2a isoprostane in serum to reflect oxidative stress. Measured at Baseline and Month 3.
Time Frame: Baseline and up to 3 months after enrollment
Population: Data unreported for participants who refused to provide blood sample
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
Number analyzed (Participants) | 2 | 4 | 7
pg/mL
  Baseline | 23144 (44504) | 10406 (27203) | 13832 (20676)
  3 months | 507 (262) | 2431 (3753) | 2580 (2667)

ADVERSE EVENTS:
Time Frame: From Baseline through the end of study, an approximate total of 3 months
Description: Per study protocol section 8, only pre-specified events and those events that are potentially related to participation in this research study must be collected.
Arm/Group | Intervention 1 (500 mg) | Intervention 2 (1000 mg) | Control (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04036110/Prot_SAP_000.pdf